CLINICAL TRIAL: NCT04977024
Title: A Phase 2 Randomized, Multi-center Study of GEO-CMO4S1 (SARS-CoV-2 Vaccine) Versus mRNA SARS-CoV-2 Vaccine in Patients Post Cellular Therapy for Hematological Malignancies
Brief Title: SARS-CoV-2 Vaccine (GEO-CM04S1) Versus mRNA SARS-COV-2 Vaccine in Patients With Blood Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GeoVax, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21163; NCI-2021-05556 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21163 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2021-06-11; First posted 2021-07-26 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: COVID-19 Infection; Hematopoietic and Lymphoid System Neoplasm; Leukemia; Lymphoma; Plasma Cell Myeloma
MeSH Terms: conditions — COVID-19; Leukemia; Lymphoma; Multiple Myeloma | interventions — COVID-19 Vaccines; COH04S1 COVID-19 vaccine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (GEO-CM04S1) (Experimental): Patients receive one dose of GEO-CM04S1 IM in the upper arm on days 0 and 28.
  Interventions: Other: Diagnostic Laboratory Biomarker Analysis; Biological: Synthetic MVA-based SARS-CoV-2 Vaccine GEO-CM04S1
- Arm II (SOC mRNA SARS-CoV-2 vaccine) (Experimental): Patients receive one dose of SOC mRNA SARS-CoV-2 vaccine IM in the upper arm on days 0 and 28.

INTERVENTIONS:
Biological: COVID-19 Vaccine — Receive SOC mRNA SARS-CoV-2 vaccine IM
Other: Diagnostic Laboratory Biomarker Analysis — Correlative studies
  Arms: Arm I (GEO-CM04S1)
Biological: Synthetic MVA-based SARS-CoV-2 Vaccine GEO-CM04S1 — Given IM
  Other Names: COH04S1; SARS-CoV-2 Vaccine COH04S1; sMVA-based SARS-CoV-2 Vaccine COH04S1; GEO-CM04S1
  Arms: Arm I (GEO-CM04S1)

SUMMARY:
This phase 2 trial studies the immune response to GEO-CM04S1 (previously designated as COH04S1) compared to standard of care (SOC) mRNA SARS-COV-2 vaccine in patients with blood cancer who have received stem cell transplant or cellular therapy.

GEO-CM04S1 belongs to a category called modified vaccinia Ankara (MVA) vaccines, created from a new version of MVA, called synthetic MVA. GEO-CM04S1 works by inducing immunity (the ability to recognize and fight against an infection) to SARS-CoV-2. The immune system is stimulated to produce antibodies against SARS-CoV-2 that would block the virus from entering healthy cells. The immune system also grows new disease fighting T cells that can recognize and destroy infected cells. Giving GEO-CM04S1 after cellular therapy may work better in reducing the chances of contracting coronavirus disease 2019 (COVID-19) or developing a severe form of COVID-19 disease in patients with blood cancer compared to SOC mRNA SARS-CoV-2 vaccine.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the biological activity and the role of timing of 2 injections of GEO-CM04S1 vaccine administered at 2.5e8 PFU/dose compared to SOC mRNA vaccine.

SECONDARY OBJECTIVES:

I. Assess safety of GEO-CM04S1 vaccine. II. Evaluation of SARS-CoV-2 S and N-specific Th1 vs Th2 polarization. III. Evaluate T-cell levels and function. IV. Evaluate activated/cycling and memory phenotype markers. V. Evaluate durability of immune responses. VI. Evaluate maintenance of immunity that can be associated with protection over the study period.

EXPLORATORY OBJECTIVE:

I. Surveillance for incidental COVID-19 infection during follow-up (1 year).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I : Patients receive one dose of GEO-CM04S1 intramuscularly (IM) in the upper arm on days 0 and 28.

ARM II : Patients receive one dose of SOC mRNA SARS-CoV-2 vaccine IM in the upper arm on days 0 and 28.

After the completion of study treatment, patients are followed up at days 7, 90, 120, 180, and 365.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant
* Age >=18 years
* Eastern Cooperative Oncology Group (ECOG) =<1
* Allogeneic or autologous hematopoietic cell transplant (HCT), cellular therapy (chimeric antigen receptor [CAR] T-cell) recipients who are at >= 3 months of infusion date of respective regimen
* Platelets >= 50,000/mm^3 (to be performed within 30 days prior to day 0 of protocol therapy unless otherwise stated)
* White blood cells (WBCs) >= 1000/mm^3 (to be performed within 30 days prior to day 0 of protocol therapy unless otherwise stated)
* Total bilirubin < 1.5 X upper limit of normal (ULN) (to be performed within 30 days prior to day 0 of protocol therapy unless otherwise stated)
* Aspartate aminotransferase (AST) < 2.5 X ULN (to be performed within 30 days prior to day 0 of protocol therapy unless otherwise stated)
* Alanine aminotransferase (ALT) < 2.5 X ULN (to be performed within 30 days prior to day 0 of protocol therapy unless otherwise stated)
* Creatinine < 1.5 X ULN (to be performed within 30 days prior to day 0 of protocol therapy unless otherwise stated)
* Negative COVID-19 PCR test
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test (to be performed within 30 days prior to day 0 of protocol therapy unless otherwise stated). If the urine pregnancy test is inconclusive a serum pregnancy test will be required
* Agreement by females and males of childbearing potential* to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 6 weeks after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 1 year (women only)

Exclusion Criteria:

* Systemic corticosteroids required for chronic conditions at doses > 0.5mg/kg/day prednisone equivalent within 7 days of enrollment
* Prior Evusheld or other anti-SARS CoV-2 prophylaxis < 2 weeks prior to enrollment
* Therapies that cause profound T-cell or B cell depletion within 30 days of enrollment
* Maintenance therapies (e.g. rituximab, Bruton tyrosine kinase inhibitors, Janus kinase inhibitors) within 30 days of enrollment
* Received investigational or licensed SARS-CoV-2 vaccines after their qualifying cellular therapy. Patients who received a SARS- CoV-2 vaccine prior to cellular therapy are eligible for this trial, as revaccination for these patients (e.g. flu and shingles vaccine) is standard of care.
* Received a live vaccine ≤30 days prior to administration of study vaccine or subjects who are =< 2 weeks within administration of inactivated vaccines (e.g. influenza vaccine). Flu shots are allowed > 2 weeks before the first injection and > 2 weeks post 2nd injection
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to vaccine agents
* History of adverse event with a prior smallpox vaccination
* Any MVA vaccine or poxvirus vaccine in the last 12 months
* History (suspected or confirmed) of myocarditis or pericarditis
* Clinically significant uncontrolled illness
* Females only: Pregnant or breastfeeding
* Any other condition that would, in the Investigator's judgment, contraindicate the subject's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)
* Anyone considered to be in a vulnerable population as defined in 45 CFR §46.111 (a)(3) and 45 CFR §46, Subparts B-D

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Biological response | At 28 days post the second vaccine injection
  Based on at least a 3-fold increase in severe acute respiratory syndrome coronavirus 2 (SARSCoV-2)- neutralizing antibodies or interferon (IFN)-gamma levels. Will compare the immune response at day 28 post the second injection between GEO-CM04S1 and SOC mRNA SARS-CoV-2 vaccine using a one-sided stratified Cochran-Mantel-Haenszel test. The point estimate and 95% confidence interval will be calculated per arm for immune response at day 28 post the second injection. Bar charts will be generated to show the immune response rate by arm overall, and by arm and strata.

SECONDARY OUTCOMES:
Incidence of moderate adverse events (AEs) | Up to 365 days
  Will assess grade 2 AEs based on Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, at least probably related to protocol treatment.
Incidence of unacceptable AEs | Up to 365 days
  Will assess grade 3-5 AEs based on CTCAE version 5.0, at least probably related to protocol treatment.
Non-relapse mortality | Up to 365 days
  Defined as death from any cause other than relapse of underlying hematologic malignancy recorded from the first injection to day 365 among all subjects.
Incidence of graft-versus-host disease (GVHD) | Up to 365 days
  Will assess the incidence of moderate/severe chronic and late-onset grade III-IV acute GVHD among allogeneic hematopoietic cell transplantation recipients only.
Incidence of Severe coronavirus disease 2019 (COVID-19) | Up to 365 days
  Will assess for confirmed COVID-19 infection with one of the following additional features from the first injection to day 365:
  * Clinical sign at rest indicative of severe systemic illness (respiratory rate >= 30 breaths per minute, heart rate >= 125 beats per minute, oxygen saturation =< 93% on room air at sea level, or partial pressure of oxygen/fraction of inspired oxygen < 300 mm Hg);
  * Respiratory failure (defined as needing high-flow oxygen, noninvasive ventilation, mechanical ventilation, or extracorporeal membrane oxygenation);
  * Evidence of shock (systolic blood pressure <90 mmHg, diastolic blood pressure < 60 mmHg, or requiring vasopressors);
  * Significant acute renal, hepatic, or neurologic dysfunction;
  * Admission to an intensive care unit;
  * Death
Th1 vs Th2 polarization | Up to 365 days
  Will evaluate SARS-CoV-2-S and -N specific Th1 (IFN gamma ng/ml) and Th2 (IL-4 ng/ml) cytokine levels following stimulation with overlapping peptide libraries specific for SARSCoV-2. Will perform dual fluorescence ELISPOT assay to detect and quantify cells secreting IFN gamma and IL-4.
Antigen specific T cell responses to the COH04S1 vaccine | Up to 365 days
  Assessed using overlapping S and N peptide libraries specific for SARS-CoV-2.
Percentages of activated/cycling and memory phenotype markers on the surface of antigen-specific T cells | Up to 365 days
  In vaccine responders, SARS-CoV-2 specific T cells will be further evaluated by measuring levels percentages of CD137 surface marker expressed on CD3+ CD8+ and CD3+ CD4+ T cells stimulated for 24 hours with either SARS-CoV-2-S or SARS-CoV-2-N overlapping peptide libraries. Will also assess the activated/cycling phenotype percentages by using the CD38, HLA-DR, Ki67 and PD1 surface markers.
Humoral immunity | Up to 365 days
  Will measure SARS-CoV-2 specific antibodies, including IgA, IgG, and IgM, in serum and saliva by enzyme linked immunosorbent assay (ELISA). Pools of SARS-CoV-2 convalescent serum or SARS-CoV-2 negative serum will be used as a positive- and negative-controls (University of California at San Diego), respectively. Antibody levels in recipients will be graphed on a time plot and compared to baseline level in donors.
Neutralizing antibodies | Up to 365 days
  Will measure and isolate the generation of neutralizing antibodies in participants, and test whether they prevent infection of a susceptible cell line with a pseudo-type of the SARS-CoV-2 virus. Evaluation of SARS-CoV-2 neutralizing antibody titers in serum samples of COH04S1 vaccinated volunteers will be performed. Will use SARS-CoV-2 lentiviral pseudovirus expressing the Spike antigen and infecting 293T cell lines engineered to express ACE2. Spike incorporation into the pseudovirus will be verified and quantified by Western blot using Spike-specific antibodies and by ELISA.

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Principal Investigator — GeoVax, Inc.
Locations (6):
- United States (6):
  - City of Hope Medical Center, Duarte, California
  - Johns Hopkins University, Baltimore, Maryland
  - U Mass Chan Medical School, Worcester, Massachusetts
  - SUNY-Stony Brook, Stony Brook, New York
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - Fred Hutchinson Cancer Center, Seattle, Washington